CLINICAL TRIAL: NCT02182817
Title: Prospective Cohort Study of Effects of Exposure to General Anaesthesia in Infancy on Neurocognitive Development
Brief Title: Exposure to General Anaesthesia in Infancy and Neurocognitive Development
Acronym: EGAIN
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: KK Women's and Children's Hospital (Other Government)
Collaborators: Institute for Human Development and Potential (IHDP), Singapore (Other)
Responsible Party: Sponsor
Other Study IDs: EGAIN 2013/552/D
Record Dates: First submitted 2014-06-10; First posted 2014-07-08 (Estimated); Last update posted 2021-02-21 (Actual); Status verified 2021-01

CONDITIONS: Central Nervous System Complications of Anesthesia; Impaired Cognition
Keywords: General Anaesthesia; Neurocognitive Development; Behaviour
MeSH Terms: conditions — Cognition Disorders; Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Buccal swabs
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- GA-Exposed Group: Exposure to general anaesthesia below 15 months of age
- Unexposed Group: Children not exposed to general anaesthesia or surgery from GUSTO cohort. (GUSTO: Growing Up Towards Healthy Outcomes in Singapore: a prospective longitudinal study providing normative data from the local population)

SUMMARY:
This prospective cohort study aims to determine if apparently healthy children with no significant co-morbidities who undergo general anaesthesia for minor surgery before 15 months of age will develop measurable deficits in neurocognitive development compared to apparently healthy children with no significant co-morbidities who do not undergo general anaesthesia or surgery.

DETAILED DESCRIPTION:
We hypothesize that healthy children exposed to general anaesthesia for minor surgery before 15 months of age will have significantly lower neurocognitive scores at 6,18, 24 and 36 months of age compared with age, and gender matched healthy children from the GUSTO cohort without prior exposure to general anaesthesia or surgery. (GUSTO: Growing Up Towards Healthy Outcomes in Singapore: a prospective longitudinal study providing normative data from the local population).

ELIGIBILITY:
Inclusion Criteria:

* Infants born > 36 weeks gestation
* No significant co-morbidities
* Who undergo general sevoflurane anaesthesia for minor surgery lasting <150 minutes (including herniotomies, orchidopexies, circumcisions and pyloromyotomies) before 15 months of age

Exclusion Criteria:

* Prematurity <36 weeks gestation
* Birth weight less than 2400g
* Presence of a genetic or chromosomal disorder
* Disorder of the central nervous system, including any seizure disorder
* Major congenital cardiac defects

Ages: 1 Day to 15 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Full-term infants with no significant co-morbidities presenting for minor surgery at KK Womens' and children's hospital, Singapore
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2013-11; Primary Completion 2019-07 (Actual); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Neurocognitive Assessment: Bayley's Scale of Infant Development-III | 24 months of age
  Bayley's Scale of Infant Development-III

SECONDARY OUTCOMES:
Neurocognitive Assessment: Deferred Imitation | 6 and 18 months of age
  Deferred imitation is used to assess declarative memory
Neurocognitive Assessment: Habituation | 6 and 18 months of age
  Determines if an infant shows 'novelty preference' when stimuli are shown repeatedly.
Behavioural Assessment: Child behaviour checklist | 24 months of age
Event Related Potential | 6 and 18 months of age
  Auditory Oddball
Visual Expectation | 6 and 18 months of age

CONTACTS AND LOCATIONS:
Overall Officials: Choon L Bong, MBChB FRCA, Principal Investigator — KK Women's and Children's Hospital
Locations (2):
- Singapore (2):
  - Singapore Institute of Clinical Sciences, Singapore
  - KK Women's and Children's Hospital. 100 Bukit Timah Road, Singapore